CLINICAL TRIAL: NCT00459069
Title: The Use of Dendritic Cell/Tumor Fusions as a Novel Tumor Vaccine in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: David Avigan, MD, Beth Israel Deaconess Medical Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-240
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Multiple Myeloma
Keywords: tumor vaccine; GM-CSF
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Dendritic Cell Tumor Fusion Vaccine — Vaccine administered on weeks 0, 3 and 6

SUMMARY:
The main purpose of this study is to test the safety of dendritic cell tumor fusion study vaccine and to determine the type and severity of any side effects associated with this study vaccine. Cancer cells have unique markers that distinguish them from normal cells of the body. These markers can potentially serve as targets for the immune system. Dendritic cells are normally found in small amounts in the body and are responsible for immune responses against "foreign" substances that enter the body. Animal studies have shown that these fused cells can stimulate powerful anti-tumor responses.

DETAILED DESCRIPTION:
* To create the study vaccine, cells will be removed from the participants tumor and fused (mixed) with powerful immune system stimulating cells (dendritic cells) obtained from the participants blood.
* Not everyone who participates in this study will be receiving the same amount of study vaccine. A small group of people will be enrolled into the study and given a certain dose. If they tolerate it well, the next group of people enrolled will receive a higher dose. This will continue until the highest dose level tolerated is determined.
* Once the screening tests are completed and it is determined the participant is eligible, they will undergo some baseline procedures. In an effort to make the study vaccine, tumor cells and dendritic cells will be collected from the participant. Tumor cells may be collected from bone marrow or from a collection of tumor cells called a plasmacytoma. A decision will be made based upon the location of the cancer.
* A bone marrow aspiration/biopsy will be performed during the following time points: at screening, prior to the first vaccination, and at 1 month, 3 months, and 6 months after the final study vaccination. These will be used to assess and follow the participants multiple myeloma.
* Leukapheresis will be performed to obtain dendritic cells. This procedure takes 2 to 4 hours to and involves the collection of a large number of white blood cells. Dendritic cells will be generated in the laboratory from white blood cells. If not enough white blood cells are collected, the participant may be asked to return to the clinic for an additional leukapheresis procedure.
* Before each vaccine is administered (weeks 0, 3, 6) the following study tests and procedures will be performed: skin test; blood test, physical exam and 24-hour urine collection. A physical exam and blood tests will be performed on the weeks when the participant does not receive the vaccine (weeks 1,2,4,5,7,8).
* The study schedule will consist of a fixed dose of the fused (mixed) cell vaccine under the skin every 3 weeks. Each study vaccine will be accompanied by an injection of GM-CSF. Participants will receive 2 or more vaccines depending upon the total number of fusion cells made, the dose the participant is assigned to receive and their response to the study vaccine.
* Follow-up after the vaccine treatment is completed will consist of the following: blood collection (1, 3 and 6 months after final study vaccination); bone marrow aspiration/biopsy (1, 3 and 6 months after final study vaccination); physical exam (1, 2, 3, 4, 5 and 6 months after final study vaccination); radiologic tumor assessment (1, 3 and 6 months after final study vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma: Stage I not requiring initiation of chemotherapy; Stage I, II or III patients felt to be clinically stable and having received at least one prior chemotherapy regimen
* Measurable disease as defined by a history of an elevated M component in plasma or urine or free kappa.lambda light chains in serum
* 18 years of age or older
* ECOG Performance Status of 0-1 with a greater than nine week life expectancy
* > 20% bone marrow involvement or plasmacytoma amenable to resection under local anesthesia
* Laboratory results within ranges outlined in protocol
* Negative pregnancy test and adequate contraception method(s) must be documented

Exclusion Criteria:

* History of clinically significant venous thromboembolism
* Received other immunotherapy treatment in the past 4 weeks prior to the initiation of cell collections for vaccine generation
* Chemotherapy or radiation therapy 4 weeks prior to the first vaccine
* Clinically significant autoimmune disease
* HIV positive
* Serious intercurrent illness
* Taking systemic corticosteroids within 4 weeks of treatment with study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-07; Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To assess the toxicity associated with vaccination of patients multiple myeloma with dendritic cell(DC)/tumor cell fusions co-administered with GM-CSF. | 5 years

SECONDARY OUTCOMES:
To determine whether evidence of tumor specific cellular and humoral immunity can be induced by serial vaccination with DC/tumor cell fusion cells co-administered with GMCSF | 5 years
to determine if vaccination with DC/tumor cell fusions co-administered with GM-CSF results in clinical disease response. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States